CLINICAL TRIAL: NCT05894278
Title: A Prescription Audit of Inpatient Department of National Accreditation Board for Hospitals and Healthcare Providers Approved Super Speciality Hospital in National Capital Region of India
Brief Title: A Prescription Audit of Inpatient Department of Super Speciality Hospital in National Capital Region of India
Status: Completed | Type: Observational
Sponsor: Kakatiya University (Other)
Collaborators: Fortis Hospital, India (Other)
Responsible Party: Principal Investigator, Satyam Suman, Department of Clinical Pharmacy and Clinical Pharmacology, Kakatiya University
Other Study IDs: FORTIS/IEC/2023/MAR/PA02
Record Dates: First submitted 2023-05-28; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Review of In-patient Prescription

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Compliance: Prescription properly filled for specific parameters
  Interventions: Other: Prescription data collection
- Non Compliance: Prescription is not filled with specific parameters
  Interventions: Other: Prescription data collection
- Not available - NA: Prescription does not contain specific data
  Interventions: Other: Prescription data collection

INTERVENTIONS:
Other: Prescription data collection — Prescription data collection

SUMMARY:
Prescription auditing is the art to check the detailing, compatibility and performance of the generated prescription from the physician to the pharmacist and patient, by means of the WHO checklist for prescription auditing. An audit is defined as the review and evaluation of the healthcare procedures and documentation to compare the quality of care provided, with accepted standards.

In this study, we will collect In-patient prescriptions from Fortis Hospital. And it will be evaluated for 13 list out parameters i.e Hospital unique ID, patient name, age, sex, weight, date of consultation, cleanliness and legibility, brief history, allergies, clinical examination, presumptive or definite diagnosis, medicine prescribed by generic name, dose, duration, history of a previous adverse event, appropriate abbreviations used, drug-drug interaction, drug duplication, doctor name, registration number and signature. The study is analyzed by Statistical Process Control (SPC).

DETAILED DESCRIPTION:
Aim of the study:

The aim of the study is to evaluate the quality of the prescription provided to the inpatient.

Objectives of the study:

To study the quality of good prescription In minimization of prescription errors and medication errors Also to comply with good clinical practice Enhancement of patient safety In the maintenance of rational prescribing To study the quality of care provided by the hospital to the patient

Plan of study:

To select the patient based on inclusion and exclusion criteria To collect the information from IP prescription and drug chart To identify prescribing errors and medication error To study the management of good prescription

Methodology:

Study Sites: Fortis Hospital, Noida, Uttar Pradesh (INDIA) Study Design: Observational cohort study Study Duration: 2 months (March, 2023 and May, 2023)

Study Sites: Fortis Hospital, Noida, Uttar Pradesh (INDIA) Study Design: Observational cohort study Study Duration: 2 months (March, 2023 and May, 2023)

Subject Eligibility:

1. Inclusion Criteria Participants who are willing to participate Participants who are admitted in the in-patient department Participants admitted during the study period Participants who have a prescription which is legible and complete
2. Exclusion Criteria Participants who are unwilling to provide the required information Participants who are not admitted the in-patient department Participants whose prescription is not legible and competent
3. Source of the data: Review of In-patient prescription

Sample Size:

300 prescriptions

ELIGIBILITY:
Inclusion Criteria:

* Participants who are willing to participate
* Participants who are admitted in the in-patient department
* Participants admitted during the study period
* Participants who have a prescription which is legible and complete

Exclusion Criteria:

* Participants who are unwilling to provide the required information
* Participants who are not admitted the in-patient department
* Participants whose prescription is not legible and competent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — No gender discrimination yet
Study Population: Select the patient based on inclusion and exclusion criteria Collect the information from IP prescription and drug chart Identify prescribing errors and medication error To study the management of good prescription
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage prescription | March 2023 and May 2023
  Prescription filled for specific parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Fortis Hospital, Noida, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No